CLINICAL TRIAL: NCT06067711
Title: Response of Liver Enzymes to 12 Weeks of Resistance Band Training Program in Burned Patients.
Brief Title: Response of Liver to 12 Weeks of Resistance Band Training Program in Burned Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Gamal Fawzy El-Sayed, Lecturer of physical therapy of surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004652
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Burns
Keywords: Plasma elevated liver enzymes
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Resistance training will be performed during 12-weeks for 3 sessions/week on non-consecutive days. The program will consist of six exercises: triceps press, biceps curl, lat pull down, leg press, leg extension and sit-ups using resistance band. Each session will last approximately 45 minutes and consist of a 5-minute warm-up with stretching following by resistance training that will be done as a cir¬cuit, ending with 5-minute cool down. The 1 repetition maximum (1RM) is measured at baseline and follow¬ing the intervention.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance band training group: (Experimental): This group includes 30 burned patients who will receive resistance training program for 12 weeks (3times/week) using resistance band in addition to their traditional physical therapy program and medical treatment.
  Interventions: Device: resistance band
- Control group: (No Intervention): This group includes 30 burned patients who will receive only their traditional physical therapy program and medical treatment.

INTERVENTIONS:
Device: resistance band — The program will consist of six exercises: triceps press, biceps curl, lat pull down, leg press, leg extension and sit-ups using resistance band.
  Arms: Resistance band training group:

SUMMARY:
Serum concentrations of alanine transaminase (ALT) and aspartate transaminase (AST) significantly increased immediately upon burn trauma and remained significantly elevated for about three years.

Resistance training has been shown to reduce the risk of insulin resistance, aminotransfer¬ase levels, dyslipidemia and impaired fasting glucose and can be beneficial for glucose-lipid metabolism.

DETAILED DESCRIPTION:
1. Measurement procedures:

   Serum blood draws will be taken by certified technicians with the participant in a seated position.

   Spectrophotometry is the measurable analysis technique using electromagnetic spectra. It deals with the ranges of wavelengths such as near ultraviolet, near-infrared and visible light. A device called a spectrophotometer is used to measure the absorbance or transmittance through a liquid sample. The spectrophotometer measures a specific wavelength and it is possible to choose any wavelength in the spectrophotometer register as the double beam sends a beam through a blank reference sample and one through the sample to be measured.

   Normal values that will be used for patients are 0-45 IU/l for Alanine transaminase (ALT) and 0-35 IU/l for Aspartate transaminase(AST) Measurements will be taken before the treatment (pre-treatment) and after 12 weeks (post-treatment).
2. Therapeutic procedures:

Resistance band for resistance training:

Resistance training will be performed for 12 weeks for 3 sessions/week on non-consecutive days. The program will consist of six exercises: triceps press, biceps curl, lat pull-down, leg press, leg extension and sit-ups using a resistance band. Each session will last approximately 45 minutes and consist of a 5-minute warm-up with stretching followed by resistance training that will be done as a cir¬cuit, ending with a 5-minute cooldown. The 1 repetition maximum (1RM) is measured at baseline and following the intervention. Initially, participants will do two circuits using 50% of their 1RM and repeat them 10 times for the first 3 weeks, progressing to two circuits, using 60% of their 1RM and repeating 10 times for the second 3 weeks. During the third 3 weeks, participants will do three circuits using 60% of their 1RM and repeat 10 times. In the last 3 weeks, patients will do three circuits using 70% of their 1RM and repeat 10 times. A 90-second rest will be allowed between sets of exercises.

ELIGIBILITY:
Inclusion Criteria:

The subject selection will be according to the following criteria:

* Age range between 20-45 years.
* Male and female patients will participate in the study.
* All patients have burn with BBSA about 30% to 50%.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Cardiac diseases.
* Burn of sole of foot.
* Exposed hand or foot tendons.
* Upper or Lower limb amputation.
* History of liver diseases.
* Body mass index (BMI=kg/cm2)<30%.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Concentration of Alanine transaminase (ALT) and Aspartate transaminase(AST) in blood plasma. | Three months
  Liver enzymes

CONTACTS AND LOCATIONS:
Overall Officials: A G Elsayed, PHD, Study Chair — Cairo University
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No